CLINICAL TRIAL: NCT03117465
Title: Based on the Method of Tract-based Spatial Statistics Investigated Scalp Acupuncture Combined Low-frequency Repetitive Transcranial Magnetic Stimulation on Brain White Matter Microstructure of Hemiplegic Patients With Stroke
Brief Title: Scalp Acupuncture Combined rTMS on Brain White Matter Microstructure of Hemiplegic Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Sixth People's Hospital (Other)
Responsible Party: Principal Investigator, Ning Zhao, Attending Physician, Shenzhen Sixth People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SZSixth_001
Record Dates: First submitted 2017-04-12; First posted 2017-04-18 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: All the hemiplegic patients were mainly derived from stroke recovery periodical inpatients from September 2015 to September 2016 in rehabilitation unit of shenzhen nanshan district people's hospital, Guangdong Province,China. All subjects were told in detail about the risks and signed informed consent before the experiment.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- the experimental group (Experimental): Stroke hemiplegia patients are randomly assigned to the experimental group (scalp acupuncture + low frequency repetitive transcranial magnetic stimulation + routine rehabilitation treatment). All patients in the day of inpatient and the fourteenth day received DTI magnetic resonance examination twice to study the change in white matter fiber microstructure.
  Interventions: Other: the experimental group
- the control group (Other): Stroke hemiplegia patients are randomly assigned to the control group (scalp acupuncture + routine rehabilitation treatment). All patients in the day of inpatient and the fourteenth day received DTI magnetic resonance examination twice to study the change in white matter fiber microstructure.
  Interventions: Other: the control group

INTERVENTIONS:
Other: the experimental group — Stroke hemiplegia patients are randomly assigned to the experimental group (scalp acupuncture + low frequency repetitive transcranial magnetic stimulation + routine rehabilitation treatment). All patients in the day of inpatient and the fourteenth day received DTI magnetic resonance examination twice to study the change in white matter fiber microstructure.
  Arms: the experimental group
Other: the control group — Stroke hemiplegia patients are randomly assigned to the control group (scalp acupuncture + routine rehabilitation treatment). All patients in the day of inpatient and the fourteenth day received DTI magnetic resonance examination twice to study the change in white matter fiber microstructure.
  Arms: the control group

SUMMARY:
To apply Bold-fMRI technology to observe and compare the differences of task-related activation of relevant brain cortex region in stroke hemiplegic patients and healthy subjects after finger grasping movement.

DETAILED DESCRIPTION:
Stroke is one of the common cerebrovascular diseases. With the improvement of medical conditions and treatment technology, the death rate of stroke patients has declined, but the disability rate has increased. In China about 50%-70% of stroke patients have the residual sequelae such as paralysis, paralalia dysfunction and so on.

Hemiplegic is the most frequent sequelae in post-stroke patients, finger movements recovery has already became the most difficult question in all the movement kinematics and dynamics rehabilitation,which affects the total movement function and ability of daily life in the patients.The finger recovery is tightly related to the neural plastic and brain function realignment.Furthermore, whether the special brain movement functional cortex area in bilateral hemispheres can be effectively activated is the crucial solved link. A number of recent literature have displayed the special brain motor area including the primary motor cortex(M1), the supplementary motor area(SMA), the premotor area(PMA), the primary sensorimotor area(SM1),the secondary area(SM2), the cingulate sulcus area(CMA) and the cerebellum hemispheres(CB). However，the study on the above-mentioned motor area synchronously activated when the patients after systematically rehabilitative treatment performed fingers grasping task was reported rarely.

Bold-fMRI technology is a new brain functional imaging technology developed on the basis of MRI in 1990s, which not only retains the anatomical imaging characteristics of ordinary MRI, but also obtains the physiological information. The emergence of Bold-fMRI technology provides a new way to study the mechanism, evaluation and prognosis of stroke rehabilitation, and it shows a good research and clinical application value in the field of rehabilitation medicine.

ELIGIBILITY:
Inclusion Criteria:

* at the same time in accordance with ischemic stroke of Chinese and western medicine diagnostic criteria;
* the first time stroke, unilateral stroke or once attack but not remnant nerve dysfunction;
* stable vital signs and clear consciousness;
* unilateral upper limb Brunnstrom evaluation;
* age from 30 to 60 years;
* the course of disease was within 1 year.

Exclusion Criteria:

* a history of epilepsy;
* the important organs function failed such as heart, lung, liver and kidney;
* serious cognitive impairment and poor compliance;
* wearing a pacemaker、intracranial metal implants, or with skull defects;
* serious cervical spine including cervical stenosis and instability of cervical spine;
* Women during pregnancy;
* patients cannot tolerate fMRI study.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-07; Primary Completion 2017-12 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Bold-fMRI examination | changes of baseline and day 14 after treatment
  To observe and compare the differences of task-related activation of relevant brain cortex region in stroke hemiplegic patients and healthy subjects after finger grasping movement.

SECONDARY OUTCOMES:
Fugl-Meyer assessment | changes of baseline and day 14 after treatment
  To evaluates and measure the motor function.

CONTACTS AND LOCATIONS:
Overall Officials: Ning Zhao, Master, Principal Investigator — Shenzhen Sixth People's Hospital

IPD SHARING:
Plan to Share IPD: Undecided